CLINICAL TRIAL: NCT01801462
Title: Simulation-based Ultrasound Training to Improve Patient Comfort and Decrease the Need for Re-examination. A Randomized Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Martin G. Tolsgaard, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-3-2012-162
Record Dates: First submitted 2013-02-23; First posted 2013-02-28 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Conditions Related to Early Pregnancy
Keywords: Medical education; Simulation; Ultrasound training; Patient safety

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simulation-based ultrasound training (Experimental): The initial training is provided on a high-fidelity Virtual-Reality (VR) simulator (Scantrainer, Medaphor). The VR simulator provides images obtained from real patients and haptic feedback from the ultrasound probe. The basic gynecologic and advanced gynecologic modules are selected for training purposes. When all modules are passed on the VR simulator, the participants receive 30 minutes of training on the low-fidelity simulator (BluePhantom) to allow participants to review the functions, they just trained, using real ultrasound equipment.
  Interventions: Other: Simulation-based training
- Control (No Intervention): Participants randomized to the control group receive traditional clinical introduction locally in the departments. This may include observation and supervised practice and the different types of clinical training provided by each department are gathered through the department's head of education and registered.

INTERVENTIONS:
Other: Simulation-based training
  Arms: Simulation-based ultrasound training

SUMMARY:
Ultrasonography has become increasingly used in many medical specialties over the last decades as smaller and less expensive ultrasound equipment has become available. Although ultrasound imaging traditionally is considered safe, its use is highly operator dependent (EFSUMB 2010). The lack of sufficient operator skills can lead to diagnostic errors that eventually compromise patient safety due to unnecessary tests or interventions (Moore & Copel 2011). A recent report from the British National Health Service (NHS) analyzed maternity claims reported to the NHS over the past decade and identified antenatal fetal ultrasound investigations as one of the four major risk areas in obstetric care (NHS 2012). This study therefore aims to explore the effects of simulation-based ultrasound training on patient comfort levels and the need for re-examination by a second physician due to diagnostic uncertainty.

DETAILED DESCRIPTION:
Background Ultrasonography has become increasingly used in many medical specialties over the last decades as smaller and less expensive ultrasound equipment has become available. Although ultrasound imaging traditionally is considered safe, its use is highly operator dependent (EFSUMB 2010). The lack of sufficient operator skills can lead to diagnostic errors that eventually compromise patient safety due to unnecessary tests or interventions (Moore & Copel 2011). A recent report from the British National Health Service (NHS) analyzed maternity claims reported to the NHS over the past decade and identified antenatal fetal ultrasound investigations as one of the four major risk areas in obstetric care (NHS 2012). Traditional ultrasound training is challenged with long learning curves and lack of standardization of competency-based training (Salvesen et al. 2010). Given the long learning curve characterizing traditional clinical training (Jang et al. 2010), proficiency in terms of independence and acceptable diagnostic accuracy may not occur during the first many months of training. Thus, some residents may not be sufficiently trained to manage independent ultrasound examinations expected from them safely. Accelerating learning curves is therefore essential from a patient safety perspective and for patient discomfort during intimate examinations such as transvaginal ultrasound scans. However, it may also be important from an organizational viewpoint as insufficiently trained residents may not be as effective in managing patients as those, who are trained until proficiency.

Simulation-based training has become increasingly used in several medical domains because it provides a safe environment to practice. Virtual Reality (VR) simulation has previously been shown to improve technical performance and shorten operation time in laparoscopic surgery (Larsen et al. 2009) and this type of training may therefore be useful as an adjunct to supervised clinical ultrasound practice. In previous studies of the effect of VR simulation, control groups have been assigned 'traditional training', which often means 'no training'. Consequently, it is not known if VR simulation - including ultrasound simulation - is superior to optimal clinical training using real patients. Furthermore, no studies have explored the effects of ultrasound simulation on patient related outcomes such as diagnostic accuracy, patient discomfort and their perception of safety during the ultrasound examinations. The effects on an organizational level such as the use of time per ultrasound examination, the need for re-examination by a senior clinician or the need for ambulatory control due to diagnostic uncertainty are also unknown.

Hence, we aim to explore the following research questions:

1) What are the effects of simulation-based training compared to traditional training in a group of OB/GYN residents without prior ultrasound experience, on the following outcomes:

1. Patients' discomfort levels and perception of safety immediately after a transvaginal ultrasound examination in a gynecological care unit.
2. Need for re-examination of the patients by a clinical supervisor after the initial examination.
3. Number of ambulatory controls needed due to diagnostic uncertainty.

Methods

Study setup In a randomized observer-blinded study, the effects of simulation-based ultrasound training compared to traditional training are examined from April 1st 2013 to January 31st 2014. Flowchart of study design is shown in Figure 3. Ethical approval is obtained from the Regional Ethical Committee of the Capital Region. The study is conducted in accordance with the Helsinki Declaration and in accordance with the CONSORT statement (www.consort-statement.org).

Participants All OB/GYN departments in eastern Denmark (Zealand) are contacted by e-mail and invited to participate in the study (N=7). Inclusion criteria require that participants 1) are medical graduates and 2) provide written informed consent. Exclusion criteria are 1) any formal ultrasound training or 2) previous independent use of ultrasound. The estimated number of eligible residents from each of the seven departments is eight during the 12 months of the study, giving a total of 56 potential participants, provided a participation rate of 100%. All participants are surveyed regarding age, years of post-graduate clinical practice, gender, handedness, and experience with video-gaming.

Randomization The Clinical Trials Unit, Rigshospitalet, independently performs simple randomization of participants by computer to either intervention group (simulation training) or control group (clinical training only). The allocation of participants is concealed to the primary investigator until all data is loaded to a database for statistical processing.

Intervention Simulation programme. Participants in the intervention group receive simulation training using two types of ultrasound simulators (see Figure 4 for flowchart of the simulation programme). A short theoretical introduction to pelvic ultrasound is presented before simulation training begins. Theoretical reading material concerning early pregnancy complications is provided all participants prior to simulation training. A final theoretical test is provided to assess knowledge about equipment, ultrasound safety, anatomical landmarks and basic pathology.

Content of simulation training. A low-fidelity simulator (BluePhantom), which allows participants to introduce the probe and familiarize themselves with the ultrasound equipment, is used for the initial training. Participants train for 30 minutes on this simulator before moving on to a high-fidelity Virtual-Reality (VR) simulator (Scantrainer, Medaphor). The VR simulator provides images obtained from real patients and haptic feedback from the ultrasound probe. The basic gynecologic and advanced gynecologic modules are selected for training purposes. The selection of modules is based on a previous pilot study, in which 10 OB/GYN residents rated the usefulness of each of the modules on the VR simulator. Only modules that are rated as four or five out of five in usefulness are included in the training programme. When all modules are passed on the VR simulator, the participants receive 30 minutes of training on the low-fidelity simulator (BluePhantom) to allow participants to review the functions, they just trained, using real ultrasound equipment.

Instructor-feedback during simulations. The participants receive 30 minutes of introduction to the VR simulator and are allowed another two times 10 minutes of instructor-feedback at a time of their choice (Østergaard et al. 2012).

Control Participants randomized to the control group receive traditional clinical introduction locally in the departments. This may include observation and supervised practice and the different types of clinical training provided by each department are gathered through the department's head of education and registered.

Follow-up and outcome All participants will be followed for six months. Patients eligible for participation are those who are having a pelvic ultrasound examination performed, are able to understand and read Danish, and willing to provide informed consent. Consenting patients are surveyed after the pelvic ultrasound examination regarding discomfort levels and perception of safety during the ultrasound examination. Both questions are answered using 10-point Likert scales. The need for re-examination by a supervising clinician, and need for ambulatory control including reason (e.g. diagnostic uncertainty, routine control according to department or national guidelines etc.) is registered by the nurse on call.

Sample size calculation A meaningful reduction in the need for a second re-examination by a senior clinician could be a 33% assuming a standard deviation of eight scans. Thus, a total sample size of 46 participants is needed using a two-sided alpha of 0.05 and a power of 0.90.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria require that participants 1) are medical graduates and 2) provide written informed consent.

Exclusion Criteria:

Exclusion criteria are 1) any formal ultrasound training or 2) previous independent use of ultrasound.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Patient comfort levels | Participants will be followed for 6 months.
  Patient comfort levels is surveyed for all patients being treated in the gynecological emergency departments.

SECONDARY OUTCOMES:
Need for re-examination of patients | 6 months
  All participants (physicians with no prior OB-GYN experience) register if they needed supervision during the ultrasound examination or if a senior gynecologists needed to perform a second ultrasound examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Juliane Marie Center, Copenhagen University Hospital Rigshospitalet, Copenhagen, Denmark